CLINICAL TRIAL: NCT03899623
Title: Multi-modal Imaging and Artificial Intelligence Diagnostic System for Multi-level Clinical Application
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, Principal Investigator, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2017KYPJ104
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Diabete Mellitus; Diabetic Retinopathy
Keywords: Diabete Mellitus; Diabetic Retinopathy; Artificial Intelligence
MeSH Terms: conditions — Diabetes Mellitus; Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is to build an multi-modal artificial intelligence ophthalmological imaging diagnostic system covering multi-level medical institutions. We are going to evaluate this system in an evidence-based medicine view, taking diabetic retinopathy as an example. And clinical diagnostic criteria will be made based on this multi-modal artificial intelligence imaging diagnostic system. The study is designed as a cross-sectional study involving 1,000 normal individuals, 1,000 diabetes patients without ocular complications, and 1,000 with diabetic ocular complications. Statistical analysis of the diagnostic sensitivity and specificity of the artificial intelligence system will be made, and ROC curve wil be draw.

ELIGIBILITY:
Inclusion Criteria:

Group A(normal individuals): Meet all the items 1 ~ 5 below

1. No familial or hereditary retinopathy;
2. No history of ocular trauma and / or history of ocular disease (except for mild to moderate refractive errors and / or age-related cataracts);
3. No drug use history that may cause side effects of retina (such as chloroquine, hydroxychloroquine, chlorpromazine, rifampin, etc.); 4 binocular diopter ≤ ± 6.00D; No systemic diseases that may affect the retina.

Group B(diabetes patients without ocular complications): meet any of 1 to 3, and both 4 to 5 items

1. Diagnosed with type 1 diabetes for more than 5 years;
2. Diagnosed with type 2 diabetes patients;
3. Diagnosis of gestational diabetes patients;
4. Without systemic disease that may affect the retina except for diabetes;
5. Meet the standards of 1 to 4 items.

Group C(patients with diabetic ocular complications): meet with any of 1 to 3, and all 4 to 6 items

1. Diagnosed with type 1 diabetes for more than 5 years;
2. Diagnosed with type 2 diabetes patients;
3. Diagnosis of gestational diabetes patients;
4. Meet the guidelines for diagnosis and treatment of diabetic retinopathy in any stage of diabetic retinopathy and / or diabetic macular edema.
5. Without systemic disease that may affect the retina except for diabetes;
6. A group to meet the criteria for 1 to 4 items.

Exclusion Criteria:

1. Refractive pathway is turbid, so that fundus image can not be clearly photographed;
2. With other fundus diseases and / or other diseases that seriously affect the visual function;
3. Any eye infection, such as conjunctivitis, keratitis, scleritis, endophthalmitis, acute and chronic dacryocystitis, or eye injury;
4. Serious systemic diseases such as diabetes, hypertension, heart failur,renal failure;
5. Can not cooperate with the examiner due to mental or other reasons.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Stratified sampling
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic sensitivity, specificity and ROC curve of the artificial intelligence（AI） system compared with reference standard (ophthalmologist). | It will take 15~20min for each subject to take the exams.
  Sensitivity: the percentage of diabetic retinopathy（DR） patients who are correctly identified as having the condition by AI. Sensitivity=True positive/(True positive+False negative). Specificity: the percentage of healthy people who are correctly identified as not having the condition by AI. Specificity=True negative /(True negative +False positive). The ROC curve was plotted with true positive rate (sensitivity) as the ordinate and false positive rate (1-specificity) as the abscissa.

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Jin, Professor, Principal Investigator — Zhongshan Opthalmic Center
Locations (1):
- Zhongshan Opthalmic Center, Guangzhou, Guangdong, China